**PROTOCOL NAME:** Epicenters for the Prevention of Healthcare Associated Infections (HAIs) -- Volume of Contamination and Nosocomial Infection Control: Specific Aim II.1 [Use of Provodine to Protect HCW Hands (Aim II.1)]

**PROTOCOL NUMBER:** 

Modification #: 0

**PROTOCOL VERSION DATE:** 10/20/2015

## **GENERAL INFORMATION**

| Name and address of the study monitor and person authorized to sign the protocol and amendments: |
|---|
| Loreen |
| UIHC Research Team: |
| Heather |
| Sandra |
| Melissa |
| Name and addresses of the study site: |
| The University of Iowa Hospitals and Clinics |
| 200 Hawkins Dr. |
| Iowa City, IA 52242 |

# **Table of Contents**

| <u>SU</u> | <u>SUMMARY</u> 4 |
|-----------|-------------------------------------------|
| 1. | BACKGROUND INFORMATION AND RATIONALE5 |
| | 1.1. BACKGROUND INFORMATION5 |
| | 1.2. <u>RATIONALE</u> 5 |
| | 1.3. <u>RISKS</u> 6 |
| | 1.4. <u>BENEFITS</u> 6 |
| | 1.5. RISK BENEFITS RATIO6 |
| 2. | STUDY OBJECTIVES6 |
| 3. | STUDY DESIGN AND PROCEDURES6 |
| 4. | SELECTION AND WITHDRAWAL OF PARTICIPANTS8 |
| | 4.1. SELECTION OF STUDY POPULATION8 |
| | 4.2. INCLUSION CRITERIA8 |
| | 4.3. EXCLUSION CRITERIA8 |
| | 4.4. PARTICIPANT WITHDRAWAL8 |
| 5. | INFORMED CONSENT PROCESS8 |
| | 5.1. RECRUITMENT |

| | 5.2. <u>ALTERATION OF CONSENT</u> | .9 |
|---|---|---|
| | 5.3. WAIVER OF HIPAA AUTHORIZATION | 9 |
| | 5.4. <u>INFORMED CONSENT PROCESS</u> ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 9 |
| 6. | STATISTICAL PLAN10 | |
| | 6.1. <u>ANALYSIS PLAN</u> | ) |
| | 6.2. <u>SAMPLE SIZE ESTIMATES</u> | .1 |
| 7. | DATA COLLECTION, HANDLING, AND STORAGE12 | |

### Summary

This study seeks to investigate whether applying Provodine<sup>TM</sup> to hands protects against self-contamination during personal protective equipment (PPE) removal.

For centuries, HCWs have used special clothing and equipment to protect themselves when caring for patients with infectious diseases. Yet, we still lack basic information about the efficacy of most PPE items, the optimal removal (doffing) procedures, and the methods for educating staff and assessing their competence.(54) Recent outbreaks of severe acute respiratory syndrome (SARS), 2009 H1N1 influenza, and Ebola highlighted these deficiencies.(1, 12, 13, 55-60) Unfortunately, lessons learned from outbreaks of SARS and 2009 H1N1 did not lead to sustained improvements in PPE designs or practices. Thus, most US hospitals had great difficulty both developing protocols for Ebola PPE use and training their staff to correctly don and doff PPE.

Participants will serve as their own controls in this pilot study, first in a control arm then a Provodine<sup>TM</sup> arm. We, the research team, will contaminate participating healthcare workers' (HCW) PPE with either bacteriophage MS2 or *S. marcescens* ATCC 14756. Participants will then doff PPE using the Centers for Disease Control's (CDC) recommended protocol. We will sample their hands using the glove juice method.(124, 125) A research assistant will monitor participants as they wash their hands with soap and water then rinse their hands with 70% ethanol. Participants will then apply Provodine<sup>TM</sup> to their hands and put on (don) fresh PPE. We will repeat the contamination, doffing, and sampling procedure.

*Hypothesis*: We hypothesize that Provodine<sup>TM</sup> will protect participants' hands from contamination with the test contaminants during PPE removal. Bacterial growth from the bag-broth cultures from the Provodine<sup>TM</sup> arm will have significantly less growth than from the control arm.

### 1 Background Information and Rationale

## 1.1 Background Information

Numerous studies have shown that HCWs' knowledge (19, 24, 61, 62) about proper use of PPE and their use of PPE (9, 10, 19, 62-68) are suboptimal. For example, Reid et al. found Canadian pediatric emergency department staff correctly identified the PPE needed for only 1 out of 6 scenarios (24). Casanova et al. noted that ~70% of simulation participants doffed PPE incorrectly despite having access to instructions from the Centers for Disease Control and Prevention (CDC); participants made errors when removing eye protection (33%-56%), N95 respirators (28%-50%), and gowns (17%).(67) In fact, few Canadian HCWs surveyed reported doing hand hygiene after removing various PPE items.(69) Moreover, only 15.4% of HCWs surveyed after the Toronto SARS outbreak reported using safe practices while caring for patients and 22.1% reported using risky practices.(65) Respondents reported being less likely to use appropriate precautions when these precautions were needed most: when caring for sicker patients (APACHE > 20) and when multiple room entries were required.(65) Furthermore, use of PPE varies by item; HCWs are more likely to wear masks, gowns, and gloves than eye protection.(62, 65, 66)

Multiple groups have assessed whether PPE prevents bacterial pathogens from contaminating the environment (70) and HCWs' clothes and bodies.(71-77) These groups demonstrated that HCWs' PPE items are often (9%-69.1%) contaminated with bacterial pathogens, including gramnegative rods (72-77), methicillin-resistant *Staphylococcus aureus* (MRSA) (75), enterococci (72), vancomycin-resistant enterococci (VRE) (73-75), multidrug resistant (MDR) *Pseudomonas aeruginosa* (PA) (76), or MDR *Acinetobacter baumannii* (AB) (76), after caring for patients and that their hands can be contaminated after they remove their gloves (0-12.7%). These investigators estimated that gloves were 77% to 100% effective in preventing hand contamination.(72, 74-76) However, Olsen et al. found glove leaks after 23.7% care episodes and only 21.9% of the participants knew their gloves were breeched.(72) Thus, HCWs often contaminate their gowns and gloves while caring for patients with resistant organisms. Furthermore, gloves, while protecting HCWs' hands, are not perfect barriers; results of the laboratory-based study by Doebbeling et al. suggest that even cleansing heavily contaminated gloves before doffing may not protect HCWs' hands from contamination.(71)

During the SARS epidemic (78) and the recent West African Ebola epidemic, HCWs were at high risk of infection.(1, 55) Data from several studies indicate that surgical masks and N95 respirators significantly decreased the risk of SARS infection among HCWs caring for patients with SARS (12, 13, 56) and that inconsistent use of PPE was associated with a higher risk of infection.(16) However, some HCWs who acquired SARS wore appropriate PPE.(18, 79-81) Some of these HCWs may have contaminated themselves during unsafe doffing or during reuse of PPE.(15, 82) Similarly, PPE is an important control measure in Ebola outbreaks (55) but some HCWs who acquired Ebola in West Africa wore PPE appropriately and may have acquired the infection through self-contamination while doffing. Investigators have found similar results for influenza.(57-60, 83-85) Despite evidence supporting PPE use, Chughtai et al. found significant variations in the policies and recommendations around mask and respirator use for protection against influenza and SARS. They postulated that these "differences may reflect the scarcity of level-one evidence.(86)" In the wake of these large and deadly viral epidemics, experts have called for new, improved PPE (87, 88) and for additional robust studies to provide data to guide practice.(89, 90)

Several groups have used fluorescent markers to assess whether HCWs contaminate themselves or the environment when they use or remove PPE.(31, 34, 91-95) Rawson et al. noted that participants' hands became contaminated when they handled the "outside of a contaminated glove" and when gloves "failed.(91)" Moreover, the type of PPE affects contamination levels. Wong et al. found that self-contamination occurred more frequently with jumpsuits than with gowns (92) and Guo et al. found that self- and environmental contamination was more frequent with plastic aprons than with disposable water resistant gowns.(93) Casanova et al. found a high rate of self-contamination (70%-100%) after HCWs doffed PPE contaminated with the bacteriophage MS2, a nonenveloped, nonpathogenic RNA virus.(96) They also found that MS2 was transferred to participants' hands more frequently (78% vs. 23%) and in higher quantity with single-gloving than with double-gloving. Double-gloving did not reduce MS2 contamination

of clothes, possibly because transmission to clothes was related to inadvertant contact with contaminated hands or gowns.(96) Like Zamora et al. (34), they noted that HCWs made more errors while removing PPE when they wore more PPE (double gloves) than when they wore less (single gloves).(67)

#### 1.2 Rationale

We did not identify any studies that assessed whether products applied to the hands could eliminate bacteria or viruses transferred to the hands from contaminated PPE either via defects in the PPE (e.g., holes in gloves) or during improper doffing. Our proposal will test Provodine<sup>TM</sup>, a unique, long-acting Povidine iodine hand rub (113), to determine whether it can eliminate organisms inoculated onto hands through glove defects or by faulty PPE doffing.

Provodine<sup>TM</sup> has a patented Amidermal® delivery platform, which allows controlled delivery of povidone iodine to the epidermis. In prior laboratory and clinical studies, Provodine<sup>TM</sup>, when applied to the skin, rapidly killed viral (influenza A H1N1, human coronavirus, feline calicivirus) and numerous bacterial pathogens (e.g., *S. aureus*, *Serratia marcescens*) (113) and continued to kill exogenous pathogens inoculated onto treated skin for at least 9 hours. Drs. Herwaldt and Diekema recently found that anesthesia providers who performed hand hygiene with Provodine<sup>TM</sup> before their first case of the day had significantly fewer bacterial colony forming units (CFU) and significantly fewer pathogens, particularly *S. aureus* and *Enterococcus sp.*, on their hands than when they performed hand hygiene with their usual hand hygiene agent (115).

#### REFERENCES:

- 1. Kilmarx PH, Clarke KR, Dietz PM, Hamel MJ, Husain F, McFadden JD, Park BJ, Sugerman DE, Bresee JS, Mermin J, McAuley J, Jambai A. Ebola virus disease in health care workers--Sierra Leone, 2014. MMWR Morb Mortal Wkly Rep. 2014;63(49):1168-71. Epub 2014/12/17. PubMed PMID: 25503921.
- 2. Pathmanathan I, O'Connor KA, Adams ML, Rao CY, Kilmarx PH, Park BJ, Mermin J, Kargbo B, Wurie AH, Clarke KR. Rapid assessment of Ebola infection prevention and control needs--six districts, Sierra Leone, October 2014. MMWR Morb Mortal Wkly Rep. 2014;63(49):1172-4. Epub 2014/12/17. PubMed PMID: 25503922.
- 3. Fischer WA, 2nd, Hynes NA, Perl TM. Protecting health care workers from Ebola: personal protective equipment is critical but is not enough. Ann Intern Med. 2014;161(10):753-4. Epub 2014/08/27. doi: 10.7326/m14-1953. PubMed PMID: 25155746.
- 4. Yap FH, Gomersall CD, Fung KS, Ho PL, Ho OM, Lam PK, Lam DT, Lyon DJ, Joynt GM. Increase in methicillin-resistant Staphylococcus aureus acquisition rate and change in pathogen pattern associated with an outbreak of severe acute respiratory syndrome. Clin Infect Dis. 2004;39(4):511-6. Epub 2004/09/10. doi: 10.1086/422641. PubMed PMID: 15356814.
- 5. Tokars JI, McKinley GF, Otten J, Woodley C, Sordillo EM, Caldwell J, Liss CM, Gilligan ME, Diem L, Onorato IM, Jarvis WR. Use and efficacy of tuberculosis infection control practices at hospitals with previous outbreaks of multidrug-resistant tuberculosis. Infect Control Hosp Epidemiol. 2001;22(7):449-55. Epub 2001/10/05. doi: 10.1086/501933. PubMed PMID: 11583215.
- 6. Menzies D, Fanning A, Yuan L, Fitzgerald M. Tuberculosis among health care workers. N Engl J Med. 1995;332(2):92-8. Epub 1995/01/12. doi: 10.1056/nejm199501123320206. PubMed PMID: 7990907.
- 7. Kellerman SE, Saiman L, San Gabriel P, Besser R, Jarvis WR. Observational study of the use of infection control interventions for Mycobacterium tuberculosis in pediatric facilities. Pediatr Infect Dis J. 2001;20(6):566-70. Epub 2001/06/23. PubMed PMID: 11419496.
- 8. Wise ME, De Perio M, Halpin J, Jhung M, Magill S, Black SR, Gerber SI, Harriman K, Rosenberg J, Borlaug G, Finelli L, Olsen SJ, Swerdlow DL, Kallen AJ. Transmission of pandemic (H1N1) 2009 influenza to healthcare personnel in the United States. Clin Infect Dis. 2011;52 Suppl 1:S198-204. Epub 2011/03/05. doi: 10.1093/cid/ciq038. PubMed PMID: 21342895.
- 9. Jaeger JL, Patel M, Dharan N, Hancock K, Meites E, Mattson C, Gladden M, Sugerman D, Doshi S, Blau D, Harriman K, Whaley M, Sun H, Ginsberg M, Kao AS, Kriner P, Lindstrom S, Jain S, Katz J, Finelli L, Olsen SJ, Kallen AJ. Transmission of 2009 pandemic influenza A (H1N1) virus among healthcare personnel-Southern California, 2009. Infect Control Hosp Epidemiol. 2011;32(12):1149-57. Epub 2011/11/15. doi: 10.1086/662709. PubMed PMID: 22080652.
- 10. Banach DB, Bielang R, Calfee DP. Factors associated with unprotected exposure to 2009 H1N1 influenza A among healthcare workers during the first wave of the pandemic. Infect Control Hosp Epidemiol. 2011;32(3):293-5. Epub 2011/04/05. doi: 10.1086/658911. PubMed PMID: 21460517.

- 11. Novel influenza A (H1N1) virus infections among health-care personnel United States, April-May 2009. MMWR Morb Mortal Wkly Rep. 2009;58(23):641-5. Epub 2009/06/23. PubMed PMID: 19543199.
- 12. Seto WH, Tsang D, Yung RW, Ching TY, Ng TK, Ho M, Ho LM, Peiris JS. Effectiveness of precautions against droplets and contact in prevention of nosocomial transmission of severe acute respiratory syndrome (SARS). Lancet. 2003;361(9368):1519-20. Epub 2003/05/10. PubMed PMID: 12737864.
- 13. Loeb M, McGeer A, Henry B, Ofner M, Rose D, Hlywka T, Levie J, McQueen J, Smith S, Moss L, Smith A, Green K, Walter SD. SARS among critical care nurses, Toronto. Emerg Infect Dis. 2004;10(2):251-5. Epub 2004/03/20. doi: 10.3201/eid1002.030838. PubMed PMID: 15030692; PubMed Central PMCID: PMCPmc3322898.
- 14. Chan-Yeung M. Severe acute respiratory syndrome (SARS) and healthcare workers. Int J Occup Environ Health. 2004;10(4):421-7. Epub 2005/02/11. doi: 10.1179/oeh.2004.10.4.421. PubMed PMID: 15702757.
- 15. Cluster of severe acute respiratory syndrome cases among protected health-care workers--Toronto, Canada, April 2003. MMWR Morb Mortal Wkly Rep. 2003;52(19):433-6. Epub 2003/06/17. PubMed PMID: 12807083.
- 16. Lau JT, Fung KS, Wong TW, Kim JH, Wong E, Chung S, Ho D, Chan LY, Lui SF, Cheng A. SARS transmission among hospital workers in Hong Kong. Emerg Infect Dis. 2004;10(2):280-6. Epub 2004/03/20. doi: 10.3201/eid1002.030534. PubMed PMID: 15030698; PubMed Central PMCID: PMCPmc3322933.
- 17. Gamage B, Moore D, Copes R, Yassi A, Bryce E. Protecting health care workers from SARS and other respiratory pathogens: a review of the infection control literature. Am J Infect Control. 2005;33(2):114-21. Epub 2005/03/12. doi: 10.1016/j.ajic.2004.12.002. PubMed PMID: 15761412.
- 18. Ofner-Agostini M, Gravel D, McDonald LC, Lem M, Sarwal S, McGeer A, Green K, Vearncombe M, Roth V, Paton S, Loeb M, Simor A. Cluster of cases of severe acute respiratory syndrome among Toronto healthcare workers after implementation of infection control precautions: a case series. Infect Control Hosp Epidemiol. 2006;27(5):473-8. Epub 2006/05/04. doi: 10.1086/504363. PubMed PMID: 16671028.
- 19. Daugherty EL, Perl TM, Needham DM, Rubinson L, Bilderback A, Rand CS. The use of personal protective equipment for control of influenza among critical care clinicians: A survey study. Crit Care Med. 2009;37(4):1210-6. Epub 2009/02/27. doi: 10.1097/CCM.0b013e31819d67b5. PubMed PMID: 19242326.
- 20. Gershon RR, Vlahov D, Felknor SA, Vesley D, Johnson PC, Delclos GL, Murphy LR. Compliance with universal precautions among health care workers at three regional hospitals. Am J Infect Control. 1995;23(4):225-36. Epub 1995/08/01. PubMed PMID: 7503434.
- 21. Gralton J, Rawlinson WD, McLaws ML. Health care workers' perceptions predicts uptake of personal protective equipment. Am J Infect Control. 2013;41(1):2-7. Epub 2012/05/29. doi: 10.1016/j.ajic.2012.01.019. PubMed PMID: 22633133.
- 22. Mitchell R, Ogunremi T, Astrakianakis G, Bryce E, Gervais R, Gravel D, Johnston L, Leduc S, Roth V, Taylor G, Vearncombe M, Weir C. Impact of the 2009 influenza A (H1N1) pandemic on Canadian health care workers: a survey on vaccination, illness, absenteeism, and personal protective equipment. Am J Infect Control. 2012;40(7):611-6. Epub 2012/05/12. doi: 10.1016/j.ajic.2012.01.011. PubMed PMID: 22575285.
- 23. Nichol K, Bigelow P, O'Brien-Pallas L, McGeer A, Manno M, Holness DL. The individual, environmental, and organizational factors that influence nurses' use of facial protection to prevent occupational transmission of communicable respiratory illness in acute care hospitals. Am J Infect Control. 2008;36(7):481-7. Epub 2008/09/13. doi: 10.1016/j.ajic.2007.12.004. PubMed PMID: 18786451.
- 24. Reid SM, Farion KJ, Suh KN, Audcent T, Barrowman NJ, Plint AC. Use of personal protective equipment in Canadian pediatric emergency departments. Cjem. 2011;13(2):71-8. Epub 2011/03/26. PubMed PMID: 21435312.
- 25. Turnberg W, Daniell W, Simpson T, Van Buren J, Seixas N, Lipkin E, Duchin J. Personal healthcare worker (HCW) and work-site characteristics that affect HCWs' use of respiratory-infection control measures in ambulatory healthcare settings. Infect Control Hosp Epidemiol. 2009;30(1):47-52. Epub 2008/12/03. doi: 10.1086/592707. PubMed PMID: 19046059.
- 26. Visentin LM, Bondy SJ, Schwartz B, Morrison LJ. Use of personal protective equipment during infectious disease outbreak and nonoutbreak conditions: a survey of emergency medical technicians. Cjem. 2009;11(1):44-56. Epub 2009/01/27. PubMed PMID: 19166639.
- 27. Weber DJ, Sickbert-Bennett EE, Brown VM, Brooks RH, Kittrell IP, Featherstone BJ, Adams TL, Rutala WA. Compliance with isolation precautions at a university hospital. Infect Control Hosp Epidemiol. 2007;28(3):358-61. Epub 2007/02/28. doi: 10.1086/510871. PubMed PMID: 17326031.
- 28. Manian FA, Ponzillo JJ. Compliance with routine use of gowns by healthcare workers (HCWs) and non-HCW visitors on entry into the rooms of patients under contact precautions. Infect Control Hosp Epidemiol. 2007;28(3):337-40. Epub 2007/02/28. doi: 10.1086/510811. PubMed PMID: 17326026.
- 29. Afif W, Huor P, Brassard P, Loo VG. Compliance with methicillin-resistant Staphylococcus aureus precautions in a teaching hospital. Am J Infect Control. 2002;30(7):430-3. Epub 2002/11/01. PubMed PMID: 12410221.
- 30. Thompson BL, Dwyer DM, Ussery XT, Denman S, Vacek P, Schwartz B. Handwashing and glove use in a long-term-care facility. Infect Control Hosp Epidemiol. 1997;18(2):97-103. Epub 1997/02/01. PubMed PMID: 9120250.
- 31. Beam EL, Gibbs SG, Boulter KC, Beckerdite ME, Smith PW. A method for evaluating health care workers' personal protective equipment technique. Am J Infect Control. 2011;39(5):415-20. Epub 2011/01/25. doi: 10.1016/j.ajic.2010.07.009. PubMed PMID: 2125874
- 32. Carrico RM, Coty MB, Goss LK, Lajoie AS. Changing health care worker behavior in relation to respiratory disease transmission with a novel training approach that uses biosimulation. Am J Infect Control. 2007;35(1):14-9. Epub 2007/02/06. doi: 10.1016/j.ajic.2005.12.013. PubMed PMID: 17276786.
- 33. Hon CY, Gamage B, Bryce EA, LoChang J, Yassi A, Maultsaid D, Yu S. Personal protective equipment in health care: can online infection control courses transfer knowledge and improve proper selection and use? Am J Infect Control. 2008;36(10):e33-7. Epub 2008/12/17. doi: 10.1016/j.ajic.2008.07.007. PubMed PMID: 19084161.
- 34. Zamora JE, Murdoch J, Simchison B, Day AG. Contamination: a comparison of 2 personal protective systems. Cmaj. 2006;175(3):249-54. Epub 2006/08/02. doi: 10.1503/cmaj.060094. PubMed PMID: 16880444; PubMed Central PMCID: PMCPmc1513425.

- 35. Muller MP, McGeer A. Febrile respiratory illness in the intensive care unit setting: an infection control perspective. Curr Opin Crit Care. 2006;12(1):37-42. Epub 2006/01/06. PubMed PMID: 16394782.
- 36. Weber DJ, Rutala WA, Schaffner W. Lessons learned: protection of healthcare workers from infectious disease risks. Crit Care Med. 2010;38(8 Suppl):S306-14. Epub 2010/08/05. doi: 10.1097/CCM.0b013e3181e69ebd. PubMed PMID: 20647788.
- 37. Fries J, Segre AM, Thomas G, Herman T, Ellingson K, Polgreen PM. Monitoring hand hygiene via human observers: how should we be sampling? Infect Control Hosp Epidemiol. 2012;33(7):689-95. Epub 2012/06/07. doi: 10.1086/666346. PubMed PMID: 22669230; PubMed Central PMCID: PMCPmc3632316.
- 38. Center UoNM. Viral Hemorrhagic Fever Donning and Doffing PPE. 2014.
- 39. Shears P, O'Dempsey TJ. Ebola virus disease in Africa: epidemiology and nosocomial transmission. J Hosp Infect. 2015;90(1):1-9. Epub 2015/02/07. doi: 10.1016/j.jhin.2015.01.002. PubMed PMID: 25655197.
- 40. Armellino D, Hussain E, Schilling ME, Senicola W, Eichorn A, Dlugacz Y, Farber BF. Using hightechnology to enforce low-technology safety measures: the use of third-party remote video auditing and realtime feedback in healthcare. Clin Infect Dis. 2012;54(1):1-7. Epub 2011/11/24. doi: 10.1093/cid/cir773. PubMed PMID: 22109950.
- 41. Armellino D, Trivedi M, Law I, Singh N, Schilling ME, Hussain E, Farber B. Replicating changes in hand hygiene in a surgical intensive care unit with remote video auditing and feedback. Am J Infect Control. 2013;41(10):925-7. Epub 2013/03/16. doi: 10.1016/j.ajic.2012.12.011. PubMed PMID: 23489740.
- 42. Zhang Z. Microsoft kinect sensor and its effect. MultiMedia, IEEE. 2012;19(2):4-10.
- 43. Han J, Shao L, Xu D, Shotton J. Enhanced computer vision with Microsoft Kinect sensor: a review. IEEE Trans Cybern.
- 2013;43(5):1318-34. Epub 2013/06/29. doi: 10.1109/tcyb.2013.2265378. PubMed PMID: 23807480.
- 44. Colagiorgio P, Romano F, Sardi F, Moraschini M, Sozzi A, Bejor M, Ricevuti G, Buizza A, Ramat S. Affordable, automatic quantitative fall risk assessment based on clinical balance scales and Kinect data. Conf Proc IEEE Eng Med Biol Soc. 2014;2014:3500-3. Epub 2015/01/09. doi: 10.1109/embc.2014.6944377. PubMed PMID: 25570745.
- 45. Gasparrini S, Cippitelli E, Spinsante S, Gambi E. A depth-based fall detection system using a Kinect(R) sensor. Sensors (Basel). 2014;14(2):2756-75. Epub 2014/02/14. doi: 10.3390/s140202756. PubMed PMID: 24521943; PubMed Central PMCID: PMCPmc3958279
- 46. Stone EE, Skubic M. Fall detection in homes of older adults using the Microsoft Kinect. IEEE J Biomed Health Inform. 2015;19(1):290-301. Epub 2014/04/16. doi: 10.1109/jbhi.2014.2312180. PubMed PMID: 24733032.
- 47. Cippitelli E, Gasparrini S, Spinsante S, Gambi E. Kinect as a tool for gait analysis: validation of a realtime joint extraction algorithm working in side view. Sensors (Basel). 2015;15(1):1417-34. Epub 2015/01/17. doi: 10.3390/s150101417. PubMed PMID: 25594588; PubMed Central PMCID: PMCPmc4327085.
- 48. Pastor I, Hayes HA, Bamberg SJ. A feasibility study of an upper limb rehabilitation system using Kinect and computer games. Conf Proc IEEE Eng Med Biol Soc. 2012;2012:1286-9. Epub 2013/02/01. doi: 10.1109/embc.2012.6346173. PubMed PMID: 23366134.
- 49. Stone EE, Butler M, McRuer A, Gray A, Marks J, Skubic M. Evaluation of the Microsoft Kinect for screening ACL injury. Conf Proc IEEE Eng Med Biol Soc. 2013:2013:4152-5. Epub 2013/10/11. doi: 10.1109/embc.2013.6610459. PubMed PMID: 24110646.
- 50. Clock SA, Cohen B, Behta M, Ross B, Larson EL. Contact precautions for multidrug-resistant organisms: Current recommendations and actual practice. Am J Infect Control. 2010;38(2):105-11. Epub 2009/11/17. doi: 10.1016/j.ajic.2009.08.008. PubMed PMID: 19913329; PubMed Central PMCID: PMCPmc2827623.
- 51. Girou E, Chai SH, Oppein F, Legrand P, Ducellier D, Cizeau F, Brun-Buisson C. Misuse of gloves: the foundation for poor compliance with hand hygiene and potential for microbial transmission? J Hosp Infect. 2004;57(2):162-9. Epub 2004/06/09. doi: 0.1016/j.jhin.2004.03.010. PubMed PMID: 15183248.
- 52. Fuller C, Savage J, Besser S, Hayward A, Cookson B, Cooper B, Stone S. "The dirty hand in the latex glove": a study of hand hygiene compliance when gloves are worn. Infect Control Hosp Epidemiol. 2011;32(12):1194-9. Epub 2011/11/15. doi: 10.1086/662619. PubMed PMID: 22080658.
- 53. Sharma D, Thomas GW, Foster ED, Iacovelli J, Lea KM, Streit JA, Polgreen PM. The precision of human-generated hand-hygiene observations: a comparison of human observation with an automated monitoring system. Infect Control Hosp Epidemiol. 2012;33(12):1259-61. Epub 2012/11/13. doi: 10.1086/668426. PubMed PMID: 23143367; PubMed Central PMCID: PMCPmc3632323
- 54. Personal Protective Equipment in the Context of Filovirus Disease Outbreak Response: Rapid Advice Guideline. 2014 [cited 05/20/2015]. Geneva: World Health Organization. Copyright (c) World Health Organization, 2014. All rights reserved.WHO Guidelines Approved by the Guidelines Review Committee, [cited 05/20/2015]. Available from: http://www.ncbi.nlm.nih.gov/books/NBK269632/pdf/TOC.pdf.
- 55. Shears P, O'Dempsey TJ. Ebola virus disease in Africa: epidemiology and nosocomial transmission. J Hosp Infect. 2015. Epub 2015/02/07. doi: 10.1016/i.jhin.2015.01.002. PubMed PMID: 25655197.
- 56. Le DH, Bloom SA, Nguyen QH, Maloney SA, Le QM, Leitmeyer KC, Bach HA, Reynolds MG, Montgomery JM, Comer JA, Horby PW, Plant AJ. Lack of SARS transmission among public hospital workers, Vietnam. Emerg Infect Dis. 2004;10(2):265-8. Epub 2004/03/20. doi: 10.3201/eid1002.030707. PubMed PMID: 15030695; PubMed Central PMCID: PMCPmc3322918.
- 57. Yeom JS, Lee JH, Bae IG, Oh WS, Moon CS, Park KH, Lee JH, Kim ES, Kwak YG, Lee CS. 2009 H1N1 influenza infection in Korean healthcare personnel. Eur J Clin Microbiol Infect Dis. 2011;30(10):1201-6. Epub 2011/03/29. doi: 10.1007/s10096-011-1213-2. PubMed PMID: 21442359.
- 58. Lee V, Yap J, Cook AR, Chen M, Tay J, Barr I, Kelso A, Tan B, Loh JP, Lin R, Cui L, Kelly PM, Leo Y, Chia K, Kang WL, Tambyah P, Seet B. Effectiveness of public health measures in mitigating pandemic influenza spread: a prospective sero-epidemiological cohort study. J Infect Dis. 2010;202(9):1319-26. Epub 2010/09/25. doi: 10.1086/656480. PubMed PMID: 20863233.
- 59. Cowling BJ, Chan KH, Fang VJ, Cheng CK, Fung RO, Wai W, Sin J, Seto WH, Yung R, Chu DW, Chiu BC, Lee PW, Chiu MC, Lee HC, Uyeki TM, Houck PM, Peiris JS, Leung GM. Facemasks and hand hygiene to prevent influenza transmission in households: a cluster randomized trial. Ann Intern Med. 2009;151(7):437-46. Epub 2009/08/05. PubMed PMID: 19652172.

- 60. Loeb M, Dafoe N, Mahony J, John M, Sarabia A, Glavin V, Webby R, Smieja M, Earn DJ, Chong S, Webb A, Walter SD. Surgical mask vs N95 respirator for preventing influenza among health care workers: a randomized trial. JAMA. 2009;302(17):1865-71. Epub 2009/10/03. doi: 10.1001/jama.2009.1466. PubMed PMID: 19797474.
- 61. Hu X, Zhang Z, Li N, Liu D, Zhang L, He W, Zhang W, Li Y, Zhu C, Zhu G, Zhang L, Xu F, Wang S, Cao X, Zhao H, Li Q, Zhang X, Lin J, Zhao S, Li C, Du B. Self-reported use of personal protective equipment among Chinese critical care clinicians during 2009 H1N1 influenza pandemic. PLoS One. 2012;7(9):e44723. Epub 2012/09/08. doi: 10.1371/journal.pone.0044723. PubMed PMID: 22957101; PubMed Central PMCID: PMCPmc3434157.
- 62. Watson CM, Duval-Arnould JM, McCrory MC, Froz S, Connors C, Perl TM, Hunt EA. Simulated pediatric resuscitation use for personal protective equipment adherence measurement and training during the 2009 influenza (H1N1) pandemic. Jt Comm J Qual Patient Saf. 2011;37(11):515-23. Epub 2011/12/03. PubMed PMID: 22132664.
- 63. Phin NF, Rylands AJ, Allan J, Edwards C, Enstone JE, Nguyen-Van-Tam JS. Personal protective equipment in an influenza pandemic: a UK simulation exercise. J Hosp Infect. 2009;71(1):15-21. Epub 2008/11/18. doi: 10.1016/j.jhin.2008.09.005. PubMed PMID: 19013670.
- 64. Parker MJ, Goldman RD. Paediatric emergency department staff perceptions of infection control measures against severe acute respiratory syndrome. Emerg Med J. 2006;23(5):349-53. Epub 2006/04/22. doi: 10.1136/emj.2005.026146. PubMed PMID: 16627834; PubMed Central PMCID: PMCPmc2564081.
- 65. Shigayeva A, Green K, Raboud JM, Henry B, Simor AE, Vearncombe M, Zoutman D, Loeb M, McGeer A. Factors associated with critical-care healthcare workers' adherence to recommended barrier precautions during the Toronto severe acute respiratory syndrome outbreak. Infect Control Hosp Epidemiol. 2007;28(11):1275-83. Epub 2007/10/11. doi: 10.1086/521661. PubMed PMID: 17926279.
- 66. Swaminathan A, Martin R, Gamon S, Aboltins C, Athan E, Braitberg G, Catton MG, Cooley L, Dwyer DE, Edmonds D, Eisen DP, Hosking K, Hughes AJ, Johnson PD, Maclean AV, O'Reilly M, Peters SE, Stuart RL, Moran R, Grayson ML. Personal protective equipment and antiviral drug use during hospitalization for suspected avian or pandemic influenza. Emerg Infect Dis. 2007;13(10):1541-7. Epub 2008/02/09. doi: 10.3201/eid1310.070033. PubMed PMID: 18258004; PubMed Central PMCID: PMCPmc2851524.
- 67. Casanova LM, Rutala WA, Weber DJ, Sobsey MD. Effect of single- versus double-gloving on virus transfer to health care workers' skin and clothing during removal of personal protective equipment. Am J Infect Control. 2012;40(4):369-74. Epub 2011/08/13. doi: 10.1016/j.ajic.2011.04.324. PubMed PMID: 21831480.
- 68. Yap FH, Ho PL, Joynt GM. Reply to Bassetti et al. Clin Infect Dis. 2005;40(4):634-5. doi: 10.1086/427155
- 69. Mitchell R, Roth V, Gravel D, Astrakianakis G, Bryce E, Forgie S, Johnston L, Taylor G, Vearncombe M. Are health care workers protected? An observational study of selection and removal of personal protective equipment in Canadian acute care hospitals. Am J Infect Control. 2013;41(3):240-4. Epub 2012/10/18. doi: 10.1016/j.ajic.2012.04.332. PubMed PMID: 23073484.
- 70. Hambraeus A. Transfer of Staphylococcus aureus via nurses' uniforms. J Hyg (Lond). 1973;71(4):799-814. Epub 1973/12/01. PubMed PMID: 4520515; PubMed Central PMCID: PMCPmc2130419.
- 71. Doebbeling BN, Pfaller MA, Houston AK, Wenzel RP. Removal of nosocomial pathogens from the contaminated glove. Implications for glove reuse and handwashing. Ann Intern Med. 1988;109(5):394-8. Epub 1988/09/01. PubMed PMID: 3136685.
- 72. Olsen RJ, Lynch P, Coyle MB, Cummings J, Bokete T, Stamm WE. Examination gloves as barriers to hand contamination in clinical practice. JAMA. 1993;270(3):350-3. Epub 1993/07/21. PubMed PMID: 8315779.
- 73. Tenorio AR, Badri SM, Sahgal NB, Hota B, Matushek M, Hayden MK, Trenholme GM, Weinstein RA. Effectiveness of gloves in the prevention of hand carriage of vancomycin-resistant enterococcus species by health care workers after patient care. Clin Infect Dis. 2001;32(5):826-9. Epub 2001/03/07. doi: 10.1086/319214. PubMed PMID: 11229854.
- 74. Hayden MK, Blom DW, Lyle EA, Moore CG, Weinstein RA. Risk of hand or glove contamination after contact with patients colonized with vancomycin-resistant enterococcus or the colonized patients' environment. Infect Control Hosp Epidemiol. 2008;29(2):149-54. Epub 2008/01/09. doi: 10.1086/524331. PubMed PMID: 18179370.
- 75. Snyder GM, Thom KA, Furuno JP, Perencevich EN, Roghmann MC, Strauss SM, Netzer G, Harris AD. Detection of methicillin-resistant Staphylococcus aureus and vancomycin-resistant enterococci on the gowns and gloves of healthcare workers. Infect Control Hosp Epidemiol. 2008;29(7):583-9. Epub 2008/06/14. doi: 10.1086/588701. PubMed PMID: 18549314; PubMed Central PMCID: PMCPmc2577846.
- 76. Morgan DJ, Liang SY, Smith CL, Johnson JK, Harris AD, Furuno JP, Thom KA, Snyder GM, Day HR, Perencevich EN. Frequent multidrug-resistant Acinetobacter baumannii contamination of gloves, gowns, and hands of healthcare workers. Infect Control Hosp Epidemiol. 2010;31(7):716-21. Epub 2010/05/22. doi: 10.1086/653201. PubMed PMID: 20486855; PubMed Central PMCID: PMCPmc3010849.
- 77. Morgan DJ, Rogawski E, Thom KA, Johnson JK, Perencevich EN, Shardell M, Leekha S, Harris AD. Transfer of multidrug-resistant bacteria to healthcare workers' gloves and gowns after patient contact increases with environmental contamination. Crit Care Med. 2012;40(4):1045-51. Epub 2011/12/29. doi: 10.1097/CCM.0b013e31823bc7c8. PubMed PMID: 22202707; PubMed Central PMCID: PMCPmc3534819.
- 78. Summary of probable SARS cases with onset of illness from 1 November 2002 to 31 July 2003 Geneva, Switzerland: World Health Organization; 2003 [updated 9/26/2003; cited 2015 5/20/2015]. Available from: http://www.who.int/csr/sars/country/table2003\_09\_23/en/.
- 79. Twu SJ, Chen TJ, Chen CJ, Olsen SJ, Lee LT, Fisk T, Hsu KH, Chang SC, Chen KT, Chiang IH, Wu YC, Wu JS, Dowell SF. Control measures for severe acute respiratory syndrome (SARS) in Taiwan. Emerg Infect Dis. 2003;9(6):718-20. Epub 2003/06/05. doi: 10.3201/eid0906.030283. PubMed PMID: 12781013; PubMed Central PMCID: PMCPmc3000163.
- 80. Mukhopadhyay A, Tambyah PA, Singh KS, Lim TK, Lee KH. SARS in a hospital visitor and her intensivist. J Hosp Infect. 2004;56(3):249-50. Epub 2004/03/09. doi: 10.1016/j.jhin.2003.12.015. PubMed PMID: 15003680.

- 81. Fowler RA, Guest CB, Lapinsky SE, Sibbald WJ, Louie M, Tang P, Simor AE, Stewart TE. Transmission of severe acute respiratory syndrome during intubation and mechanical ventilation. Am J Respir Crit Care Med. 2004;169(11):1198-202. Epub 2004/03/03. doi: 10.1164/rccm.200305-715OC. PubMed PMID: 14990393.
- 82. Shaw K. The 2003 SARS outbreak and its impact on infection control practices. Public Health. 2006;120(1):8-14. Epub 2005/11/22. doi: 10.1016/j.puhe.2005.10.002. PubMed PMID: 16297415.
- 83. Marshall C, Kelso A, McBryde E, Barr IG, Eisen DP, Sasadeusz J, Buising K, Cheng AC, Johnson P, Richards M. Pandemic (H1N1) 2009 risk for frontline health care workers. Emerg Infect Dis. 2011;17(6):1000-6. Epub 2011/07/14. doi: 10.3201/eid/1706.101030. PubMed PMID: 21749760; PubMed Central PMCID: PMCPmc3358191.
- 84. MacIntyre CR, Seale H, Dung TC, Hien NT, Nga PT, Chughtai AA, Rahman B, Dwyer DE, Wang Q. A cluster randomised trial of cloth masks compared with medical masks in healthcare workers. BMJ Open. 2015;5(4):e006577. Epub 2015/04/24. doi:
- 10.1136/bmjopen-2014-006577. PubMed PMID: 25903751; PubMed Central PMCID: PMCPmc4420971.
- 85. MacIntyre CR, Wang Q, Cauchemez S, Seale H, Dwyer DE, Yang P, Shi W, Gao Z, Pang X, Zhang Y, Wang X, Duan W, Rahman B, Ferguson N. A cluster randomized clinical trial comparing fit-tested and non-fittested N95 respirators to medical masks to prevent respiratory virus infection in health care workers. Influenza Other Respir Viruses. 2011;5(3):170-9. Epub 2011/04/12. doi: 10.1111/j.1750-2659.2011.00198.x. PubMed PMID: 21477136.
- 86. Chughtai AA, Seale H, MacIntyre CR. Availability, consistency and evidence-base of policies and guidelines on the use of mask and respirator to protect hospital health care workers: a global analysis. BMC Res Notes. 2013;6:216. Epub 2013/06/04. doi: 10.1186/1756-0500-6-216. PubMed PMID: 23725338; PubMed Central PMCID: PMCPmc3693993.
- 87. Edmond MB, Diekema DJ, Perencevich EN. Ebola virus disease and the need for new personal protective equipment. JAMA. 2014;312(23):2495-6. Epub 2014/10/29. doi: 10.1001/jama.2014.15497. PubMed PMID: 25350321.
- 88. Sprecher AG, Caluwaerts A, Draper M, Feldmann H, Frey CP, Funk RH, Kobinger G, Le Duc JW, Spiropoulou C, Williams WJ. Personal Protective Equipment for Filovirus Epidemics: A Call for Better Evidence. J Infect Dis. 2015. Epub 2015/03/31. doi: 10.1093/infdis/jiv153. PubMed PMID: 25821225.
- 89. Srinivasan A, Perl TM. Respiratory protection against influenza. Jama. 2009;302(17):1903-4. Epub 2009/10/03. doi: 10.1001/jama.2009.1494. PubMed PMID: 19797473.
- 90. Verbeek J, Ijaz S, Mischke C, Ruotsalainen J, Mäkelä E, Neuvonen K, Edmond M, Garne rP, Sauni R, Hopping K. Personal protective equipment for preventing highly infectious diseases due to contact with contaminated body fluids in health care staff (protocol). Cochrane Database Syst Rev. 2015(4). doi: 10.1002/14651858.CD011621.
- 91. Rawson BV, Cocker J, Evans PG, Wheeler JP, Akrill PM. Internal contamination of gloves: routes and consequences. Ann Occup Hyg. 2005;49(6):535-41. Epub 2005/05/19. doi: 10.1093/annhyg/mei015. PubMed PMID: 15899931.
- 92. Wong TK, Chung JW, Li Y, Chan WF, Ching PT, Lam CH, Chow CB, Seto WH. Effective personal protective clothing for health care workers attending patients with severe acute respiratory syndrome. Am J Infect Control. 2004;32(2):90-6. Epub 2004/04/02. doi: 10.1016/j.ajic.2003.08.004. PubMed PMID: 15057200.
- 93. Guo YP, Li Y, Wong PL. Environment and body contamination: a comparison of two different removal methods in three types of personal protective clothing. Am J Infect Control. 2014;42(4):e39-45. Epub 2014/04/01. doi: 10.1016/j.ajic.2013.12.021. PubMed PMID: 24679582.
- 94. Beam EL, Gibbs SG, Hewlett AL, Iwen PC, Nuss SL, Smith PW. Method for investigating nursing behaviors related to isolation care. Am J Infect Control. 2014;42(11):1152-6. Epub 2014/12/03. doi: 10.1016/j.ajic.2014.08.001. PubMed PMID: 25444261.
- 95. Tomas M, Kundrapu S, Thota P, Sunkesula V, Cadnum J, Mana T, Jencson A, Hecker M, Ray A, Donskey C. Frequent Contamination of the Skin and Clothing of Healthcare Personnel during Removal of Personal Protective Equipment: A Multicenter Evaluation and Educational Intervention. SHEA Spring 2015: Science Guiding Prevention; Orlando, Florida, 2015.
- 96. Casanova L, Alfano-Sobsey E, Rutala WA, Weber DJ, Sobsey M. Virus transfer from personal protective equipment to healthcare employees' skin and clothing. Emerg Infect Dis. 008;14(8):1291-3. Epub 2008/08/06. doi: 10.3201/eid1408.080085. PubMed PMID: 18680659; PubMed Central PMCID: PMCPmc2600382.
- 97. Nicol PW, Watkins RE, Donovan RJ, Wynaden D, Cadwallader H. The power of vivid experience in hand hygiene compliance. J Hosp Infect. 2009;72(1):36-42. Epub 2009/03/14. doi: 10.1016/j.jhin.2009.01.021. PubMed PMID: 19282058.
- 98. Widmer AF, Conzelmann M, Tomic M, Frei R, Stranden AM. Introducing alcohol-based hand rub for hand hygiene: the critical need for training. Infect Control Hosp Epidemiol. 2007;28(1):50-4. Epub 2007/01/19. doi: 10.1086/510788. PubMed PMID: 17230387.
- 99. Neves HC, Souza AC, Medeiros M, Munari DB, Ribeiro LC, Tipple AF. Safety of nursing staff and determinants of adherence to personal protective equipment. Rev Lat Am Enfermagem. 2011;19(2):354-61. Epub 2011/05/18. PubMed PMID: 21584383.
- 100. Havenith G, Heus R. A test battery related to ergonomics of protective clothing. Appl Ergon. 2004;35(1):3-20. Epub 2004/02/27. doi: 10.1016/j.apergo.2003.11.001. PubMed PMID: 14985136.
- 101. Larson EL, Liverman CT. Designing and Engineering Effective PPE 2011. Available from:
- http://www.ncbi.nlm.nih.gov/books/NBK209586/.
- 102. Williams CK. An Assessment Tool and Interactive Simulation for Using Healthcare Personal Protective Equipment. Toronto, Ontario, Canada: University of Toronto; 2010.
- 103. Davis J, Authority PPS. Equipment, Environment, and Ergonomics: An Enigma of Infection Risk. Pa Patient Saf Advis. 2015;12:37-40.
- 104. Keebler J, Gurses A, Cafazzo J, DiazGranados D, Doyle S, Feldman M, Misari P, Yazdi Y, editors. Combating Ebola: The Role of HF/E Response to the Recent EVD Outbreak. Discussion Panel. . 2015 International Symposium on Human Factors and Ergonomics in Health Care: Improving the Outcomes; 2015; Baltimore, Maryland, .
- 105. Alexander BM. Contamination of Firefighter Personal Protective Gear. Cincinnati, OH: University of Cincinnati; 2012.
- 106. Coca A, Roberge R, Shepherd A, Powell JB, Stull JO, Williams WJ. Ergonomic comparison of a chem/bio prototype firefighter ensemble and a standard ensemble. Eur J Appl Physiol. 2008;104(2):351-9. Epub 2007/12/14. doi: 10.1007/s00421-007-0644-z. PubMed PMID: 18075754.

- 107. Coca A, Williams WJ, Roberge RJ, Powell JB. Effects of fire fighter protective ensembles on mobility and performance. Appl Ergon. 2010;41(4):636-41. Epub 2010/02/16. doi: 10.1016/j.apergo.2010.01.001. PubMed PMID: 20153458.
- 108. Elder S, Hennessy E, Kanagaki G. Ergonomics evaluation of law enforcement chemical/biological (CB) personal protective equipment for the law enforcement advanced protection (LEAP) CB standards assessment. DTIC Document, 2010.
- 109. Blacker SD, Carter JM, Wilkinson DM, Richmond VL, Rayson MP, Peattie M. Physiological responses of Police Officers during job simulations wearing chemical, biological, radiological and nuclear personal protective equipment. Ergonomics. 2013;56(1):137-47. Epub 2012/11/13. doi: 10.1080/00140139.2012.734335. PubMed PMID: 23140326.
- 110. Moore D, Gamage B, Bryce E, Copes R, Yassi A. Protecting health care workers from SARS and other respiratory pathogens: organizational and individual factors that affect adherence to infection control guidelines. Am J Infect Control. 2005;33(2):88-96. Epub 2005/03/12. doi: 10.1016/j.ajic.2004.11.003. PubMed PMID: 15761408.
- 111. Lai JY, Guo YP, Or PP, Li Y. Comparison of hand contamination rates and environmental contamination levels between two different glove removal methods and distances. Am J Infect Control. 2011;39(2):104-11. Epub 2010/09/28. doi: 10.1016/j.ajic.2010.06.007. PubMed PMID: 20869790.
- 112. Hung PP, Choi KS, Chiang VC. Using interactive computer simulation for teaching the proper use of personal protective equipment. Comput Inform Nurs. 2015;33(2):49-57. Epub 2014/12/19. doi: 10.1097/cin.0000000000000125. PubMed PMID: 25521788.
- 113. MicroDermis (www.microdermis.com). ProvodineTM Investigator's Brochure. 2013.
- 114. Wigglesworth-Ballard L. A Study of a Simulated Infectious Disease on Healthcare Workers' Reaction, Knowledge, Attitudes, and Performance Towards Hand Hygiene (Unpublished doctoral dissertation). 2015.
- 115. Herwaldt L, Ford B, Chiang H-Y, Cobb S, Diekema D, Heilmann K, Jacobs P, Manning A, Riahi F, Stringham S, Todd M, Reddy S. Efficacy of ProvodineTM in Preventing Contamination of Anesthesia Providers' Hands during General Anesthesia Procedures. Interscience Conference of Antimicrobial Agents and Chemotherapy (ICAAC); 9/05/2014-9/09/2015; Washington, District of Columbia, 2014.
- 116. Wigglesworth-Ballard L. Improving nursing infection control practices in a virtual intensive care unit. Modeling, Simulation & Visualization Student Capstone Conference: Final Proceedings; Old Dominion University, Norfolk, VA, 2011. Available from: http://www.vmasc.odu.edu/downloads/CAPSTONE2011Final\_Proceedings.pdf. p. 185-90.
- 117. Moeckli J, Cram P, Cunningham C, Reisinger HS. Staff acceptance of a telemedicine intensive care unit program: a qualitative study. J Crit Care. 2013;28(6):890-901. Epub 2013/08/03. doi: 10.1016/j.jcrc.2013.05.008. PubMed PMID: 23906904.
- 118. Buzza C, Ono SS, Turvey C, Wittrock S, Noble M, Reddy G, Kaboli PJ, Reisinger HS. Distance is relative: unpacking a principal barrier in rural healthcare. J Gen Intern Med. 2011;26 Suppl 2:648-54. Epub 2011/10/19. doi: 10.1007/s11606-011-1762-1. PubMed PMID: 21989617; PubMed Central PMCID: PMCPmc3191222.
- 119. Reisinger HS. Counting apples as oranges: epidemiology and ethnography in adolescent substance abuse treatment. Qual Health Res. 2004;14(2):241-58. Epub 2004/02/11. doi: 10.1177/1049732303260670. PubMed PMID: 14768460.
- 120. Reisinger HS, Schwartz RP, Mitchell SG, Peterson JA, Kelly SM, O'Grady KE, Marrari EA, Brown BS, Agar MH. Premature discharge from methadone treatment: patient perspectives. J Psychoactive Drugs. 2009;41(3):285-96. Epub 2009/12/17. doi: 0.1080/02791072.2009.10400539. PubMed PMID: 19999682; PubMed Central PMCID: PMCPmc2796585.
- 121. Reisinger HS, Perencevich EN, Morgan DJ, Forrest GN, Shardell M, Schweizer ML, Graham MM, Franciscus CL, Vander Weg MW. Improving hand hygiene compliance with point-of-use reminder signs designed using theoretically grounded messages. Infect Control Hosp Epidemiol. 2014;35(5):593-4. Epub 2014/04/09. doi: 10.1086/675827. PubMed PMID: 24709734.
- 122. Yin J, Reisinger HS, Vander Weg M, Schweizer ML, Jesson A, Morgan DJ, Forrest G, Graham M, Pineles L, Perencevich EN. Establishing evidence-based criteria for directly observed hand hygiene compliance monitoring programs: a prospective, multicenter cohort study. Infect Control Hosp Epidemiol. 2014;35(9):1163-8. Epub 2014/08/12. doi: 10.1086/677629. PubMed PMID: 25111925. 123. Jones MV, Bellamy K, Alcock R, Hudson R. The use of bacteriophage MS2 as a model system to evaluate virucidal hand disinfectants. J Hosp Infect. 1991;17(4):279-85. Epub 1991/04/01. PubMed PMID: 1677653.
- 124. ASTM E2755-10. Standard Test Method for Determining the Bacteria-Eliminating Effectiveness of Hand Sanitizer Formulations Using Hands of Adults. West Conshohocken, PA: ASTM International; 2010.
- 125. ASTM E2011-13. Standard Test Method for Evaluation of Hygienic Handwash and Handrub
- Formulations for Virus-Eliminating Activity Using the Entire Hand. West Conshohocken, PA: ASTM International; 2013.
- 126. Environmenal Protection Agency. Method 1601: male-specific (F+) and somatic coliphage in water by two-step enrichment procedure. 2001. Available from http://www.epa.gov/nerlcwww/documents/1601ap01.pdf.
- 127. ASTM E1174-06. Standard Test Method for Evaluation of the Effectiveness of Health Care Personnel or Consumer Handwash Formulations. West Conshohocken, PA: ASTM International; 2006.
- 128. Stanton NA, Walker GH. Human factors methods: a practical guide for engineering and design: Ashgate Publishing, Ltd.; 2013.
- $129.\ Wickens\ CD,\ Gordon\ SE,\ Liu\ Y.\ An\ introduction\ to\ human\ factors\ engineering.\ 2004.$
- 130. Kirwan B, Ainsworth LK. A guide to task analysis: the task analysis working group: CRC press; 1992.
- 131. Schraagen JM, Chipman SF, Shalin VL. Cognitive task analysis: Psychology Press; 2000.
- 132. Crandall B, Klein GA, Hoffman RR. Working minds: A practitioner's guide to cognitive task analysis: Mit Press; 2006.
- 133. Goldberg JH, Wichansky AM. Eye tracking in usability evaluation: A practitioner's guide. To appear in: Hyönä. 2002.
- 134. Dixon-Woods M, Leslie M, Bion J, Tarrant C. What counts? An ethnographic study of infection data reported to a patient safety program. Milbank Q. 2012;90(3):548-91. Epub 2012/09/19. doi: 10.1111/j.1468-0009.2012.00674.x. PubMed PMID: 22985281; PubMed Central PMCID: PMCPmc3479383.
- 135. Williams CK, Carnahan H. Development and validation of tools for assessing use of personal protective equipment in health care. Am J Infect Control. 2013;41(1):28-32. Epub 2012/06/19. doi: 10.1016/j.ajic.2012.01.027. PubMed PMID: 22704736.
- 136. Ericcson K, Simon H. Protocol analysis: Verbal reports as data (revised ed.). Cambridge: MIT Press; 1996.
- 137. Krahmer E, Ummelen N. Thinking about thinking aloud: A comparison of two verbal protocols for usability testing. Professional Communication, IEEE Transactions on. 2004;47(2):105-17.

- 138. Van Den Haak M, De Jong M, Jan Schellens P. Retrospective vs. concurrent think-aloud protocols: testing the usability of an online library catalogue. Behaviour & Information Technology. 2003;22(5):339-51.
- 139. Van den Haak MJ, de Jong MD, editors. Exploring two methods of usability testing: concurrent versus retrospective think-aloud protocols. Professional Communication Conference, 2003 IPCC 2003 Proceedings IEEE International; 2003: IEEE.
- 140. Maughan L, Dodd J, Walters R. Video replay of eye tracking as a cue in retrospective protocol...don't make me think aloud! Scandinavian Workshop of Applied Eye Tracking2003.
- 141. Hyrskykari A, Ovaska S, Majaranta P, Räihä K-J, Lehtinen M. Gaze path stimulation in retrospective think-aloud. Journal of Eye Movement Research. 2008;2(4):1-18.
- 142. Weinstein RA. Epidemiology and control of nosocomial infections in adult intensive care units. Am J Med. 1991;91(3B):179S-84S. PubMed PMID: 1928162.
- 143. Samore MH, Venkataraman L, DeGirolami PC, Arbeit RD, Karchmer AW. Clinical and molecular epidemiology of sporadic and clustered cases of nosocomial Clostridium difficile diarrhea. Am J Med. 1996;100(1):32-40. PubMed PMID: 8579084.
- 144. Anderson DJ, Gergen MF, Smathers E, Sexton DJ, Chen LF, Weber DJ, Rutala WA. Decontamination of targeted pathogens from patient rooms using an automated ultraviolet-C-emitting device. Infect Control Hosp Epidemiol. 2013;34(5):466-71. doi: 10.1086/670215. PubMed PMID: 23571362; PubMed Central PMCID: PMC3703853.
- 145. Passaretti CL, Otter JA, Reich NG, Myers J, Shepard J, Ross T, Carroll KC, Lipsett P, Perl TM. An evaluation of environmental decontamination with hydrogen peroxide vapor for reducing the risk of patient acquisition of multidrug-resistant organisms. Clin Infect Dis. 2013;56(1):27-35. doi: 10.1093/cid/cis839. PubMed PMID: 23042972.
- 146. Salgado CD, Sepkowitz KA, John JF, Cantey JR, Attaway HH, Freeman KD, Sharpe PA, Michels HT, Schmidt MG. Copper surfaces reduce the rate of healthcare-acquired infections in the intensive care unit. Infect Control Hosp Epidemiol. 2013;34(5):479-86. doi: 10.1086/670207. PubMed PMID: 23571364.
- 147. Schweizer M, Graham M, Ohl M, Heilmann K, Boyken L, Diekema D. Novel hospital curtains with antimicrobial properties: a randomized, controlled trial. Infect Control Hosp Epidemiol. 2012;33(11):1081-5. doi: 10.1086/668022. PubMed PMID: 23041804. 148. Best EL, Sandoe JA, Wilcox MH. Potential for aerosolization of Clostridium difficile after flushing toilets: the role of toilet lids in reducing environmental contamination risk. J Hosp Infect. 2012;80(1):1-5. doi: 10.1016/j.jhin.2011.08.010. PubMed PMID: 22137761.
- 149. Monette M. Flush and run. CMAJ. 2012;184(11):E581-2. doi: 10.1503/cmaj.109-4196. PubMed PMID: 22761477; PubMed Central PMCID: PMC3414618.
- 150. Johnson DL, Mead KR, Lynch RA, Hirst DV. Lifting the lid on toilet plume aerosol: a literature review with suggestions for future research. Am J Infect Control. 2013;41(3):254-8. doi: 10.1016/j.ajic.2012.04.330. PubMed PMID: 23040490.
- 151. Del Rio C, Mehta AK, Lyon GM, 3rd, Guarner J. Ebola hemorrhagic fever in 2014: the tale of an evolving epidemic. Ann Intern Med. 2014;161(10):746-8. doi: 10.7326/M14-1880. PubMed PMID: 25133433.
- 152. Rock C, Thom KA, Masnick M, Johnson JK, Harris AD, Morgan DJ. Frequency of Klebsiella pneumoniae carbapenemase (KPC)-producing and non-KPC-producing Klebsiella species contamination of healthcare workers and the environment. Infect Control Hosp Epidemiol. 2014;35(4):426-9. doi: 10.1086/675598. PubMed PMID: 24602950; PubMed Central PMCID: PMC4030386.
- 153. Johnson D, Lynch R, Marshall C, Mead K, Hirst D. Aerosol Generation by Modern Flush Toilets. Aerosol Science and Technology. 2013;47(9):1047-57. doi: 10.1080/02786826.2013.814911. PubMed PMID: WOS:000324725700011.
- 154. Barker J, Jones MV. The potential spread of infection caused by aerosol contamination of surfaces after flushing a domestic toilet. J Appl Microbiol. 2005;99(2):339-47. doi: 10.1111/j.1365-2672.2005.02610.x. PubMed PMID: 16033465.
- 155. Faires MC, Pearl DL, Berke O, Reid-Smith RJ, Weese JS. The identification and epidemiology of meticillin-resistant Staphylococcus aureus and Clostridium difficile in patient rooms and the ward environment. BMC Infect Dis. 2013;13:342. Epub 2013/07/26. doi: 10.1186/1471-2334-13-342. PubMed PMID: 23883171; PubMed Central PMCID: PMC3727943.
- 156. Shaughnessy MK, Micielli RL, DePestel DD, Arndt J, Strachan CL, Welch KB, Chenoweth CE. Evaluation of hospital room assignment and acquisition of Clostridium difficile infection. Infect Control Hosp Epidemiol. 2011;32(3):201-6. doi: 10.1086/658669. PubMed PMID: 21460503.
- 157. Chang VT, Nelson K. The role of physical proximity in nosocomial diarrhea. Clin Infect Dis. 2000;31(3):717-22. Epub 2000/10/06. doi: 10.1086/314030. PubMed PMID: 11017821.
- 158. Dubberke ER, Reske KA, Olsen MA, McMullen KM, Mayfield JL, McDonald LC, Fraser VJ. Evaluation of Clostridium difficile-associated disease pressure as a risk factor for C difficile-associated disease. Arch Intern Med. 2007;167(10):1092-7. Epub 2007/05/30. doi: 10.1001/archinte.167.10.1092. PubMed PMID: 17533213.
- 159. Huang SS, Datta R, Platt R. Risk of acquiring antibiotic-resistant bacteria from prior room occupants. Arch Intern Med. 2006;166(18):1945-51. Epub 2006/10/13. doi: 10.1001/archinte.166.18.1945. PubMed PMID: 17030826.
- 160. Kramer A, Schwebke I, Kampf G. How long do nosocomial pathogens persist on inanimate surfaces? A systematic review. BMC Infect Dis. 2006;6:130. doi: 10.1186/1471-2334-6-130. PubMed PMID: 16914034; PubMed Central PMCID: PMC1564025.
- 161. Perencevich EN, Lautenbach E. Infection prevention and comparative effectiveness research. JAMA. 2011;305(14):1482-3. doi: 10.1001/jama.2011.450. PubMed PMID: 21486981.
- 162. Platt R, Takvorian SU, Septimus E, Hickok J, Moody J, Perlin J, Jernigan JA, Kleinman K, Huang SS. Cluster randomized trials in comparative effectiveness research: randomizing hospitals to test methods for prevention of healthcare-associated infections. Med Care. 2010;48(6 Suppl):S52-7. Epub 2010/05/18. doi: 10.1097/MLR.0b013e3181dbebcf. PubMed PMID: 20473200.
- 163. Cook TD, Shadish WR, Wong VC. Three conditions under which experiments and observational studies produce comparable causal estimates: New findings from within-study comparisons. Journal of Policy Analysis and Management. 2008;27(4):724-50. doi: 10.1002/pam.20375.
- 164. Harris AD, Pineles L, Belton B, Johnson JK, Shardell M, Loeb M, Newhouse R, Dembry L, Braun B, Perencevich EN, Hall KK, Morgan DJ, Benefits of Universal G, Gown I, Shahryar SK, Price CS, Gadbaw JJ, Drees M, Kett DH, Munoz-Price LS, Jacob JT, Herwaldt LA, Sulis CA, Yokoe DS, Maragakis L, Lissauer ME, Zervos MJ, Warren DK, Carver RL, Anderson DJ, Calfee DP, Bowling JE, Safdar N.

- Universal glove and gown use and acquisition of antibiotic-resistant bacteria in the ICU: a randomized trial. JAMA.
- 2013;310(15):1571-80. doi: 10.1001/jama.2013.277815. PubMed PMID: 24097234; PubMed Central PMCID: PMC4026208.
- 165. Evans ME, Simbartl LA, Kralovic SM, Jain R, Roselle GA. Clostridium difficile infections in Veterans Health Administration acute care facilities. Infect Control Hosp Epidemiol. 2014;35(8):1037-42. doi: 10.1086/677151. PubMed PMID: 25026621.
- 166. National Healthcare Safety Network (NHSN): Centers for Disease Control and Prevention; [cited 2015 May 20]. Available from: http://www.cdc.gov/nhsn/.
- 167. Methicillin-resistant Staphylococcus aureus (MRSA) prevention initiative. Directive 2010–006: Veterans Health Administration; 2010. Available from: http://www.va.gov/vhapublications/ViewPublication.asp?pub ID=2163.
- 168. Goto M, Ohl ME, Schweizer ML, Perencevich EN. Accuracy of administrative code data for the surveillance of healthcare-associated infections: a systematic review and meta-analysis. Clin Infect Dis. 2014;58(5):688-96. doi: 10.1093/cid/cit737. PubMed PMID: 24218103.
- 169. Thompson SG, Pyke SD, Hardy RJ. The design and analysis of paired cluster randomized trials: an application of meta-analysis techniques. Stat Med. 1997;16(18):2063-79. Epub 1997/10/06. PubMed PMID: 9308132.
- 170. Evans CT, Safdar N. Current Trends in the Epidemiology and Outcomes of Clostridium difficile Infection. Clin Infect Dis. 2015;60 Suppl 2:S66-71. Epub 2015/04/30. doi: 10.1093/cid/civ140. PubMed PMID: 25922403.
- 171. Ohl M, Schweizer M, Graham M, Heilmann K, Boyken L, Diekema D. Hospital privacy curtains are frequently and rapidly contaminated with potentially pathogenic bacteria. Am J Infect Control. 2012;40(10):904-6. doi: 10.1016/j.ajic.2011.12.017. PubMed PMID: 22464039.
- 172. de Smet AM, Kluytmans JA, Blok HE, Mascini EM, Benus RF, Bernards AT, Kuijper EJ, Leverstein-van Hall MA, Jansz AR, de Jongh BM, van Asselt GJ, Frenay IH, Thijsen SF, Conijn SN, Kaan JA, Arends JP, Sturm PD, Bootsma MC, Bonten MJ. Selective digestive tract decontamination and selective oropharyngeal decontamination and antibiotic resistance in patients in intensive-care units: an open-label, clustered group randomised, crossover study. Lancet Infect Dis. 2011;11(5):372-80. doi: 10.1016/S1473-3099(11)70035-4. PubMed PMID: 21420908.
- 173. Jensen PA, Schafer MP. Sampling and characterization of bioaerosols. NIOSH manual of analytical methods. 1998;1(15):82-112. 174. Dillon HK, Heinsohn PA, Miller JD. Field guide for the determination of biological contaminants in environmental samples: AIHA; 2005.
- 175. Tang CS, Chung FF, Lin MC, Wan GH. Impact of patient visiting activities on indoor climate in a medical intensive care unit: a 1-year longitudinal study. Am J Infect Control. 2009;37(3):183-8. doi: 10.1016/j.ajic.2008.06.011. PubMed PMID: 19178985.
- 176. Tang CS, Wan GH. Air quality monitoring of the post-operative recovery room and locations surrounding operating theaters in a medical center in Taiwan. PLoS One. 2013;8(4):e61093. doi: 10.1371/journal.pone.0061093. PubMed PMID: 23573296; PubMed Central PMCID: PMC3616048.
- 177. Pfaller M, Caliendo A, Versalovic J. Chromosomal restriction fragment analysis by pulsed-field gel electrophoresis: Application to molecular epidemiology. In: Garcia L, editor. Clinical Microbiology Procedures Handbook. Washington, DC: ASM Press; 2010. p. 12.4.5.1-4.5.7.
- 178. Wenzel RP, Edmond MB. Infection control: the case for horizontal rather than vertical interventional programs. Int J Infect Dis. 2010;14 Suppl 4:S3-5. doi: 10.1016/j.ijid.2010.05.002. PubMed PMID: 20851010.
- 179. Yin J, Schweizer ML, Herwaldt LA, Pottinger JM, Perencevich EN. Benefits of universal gloving on hospital-acquired infections in acute care pediatric units. Pediatrics. 2013;131(5):e1515-20. doi: 10.1542/peds.2012-3389. PubMed PMID: 23610206.
- 180. Wright MO, Hebden JN, Harris AD, Shanholtz CB, Standiford HC, Furuno JP, Perencevich EN. Aggressive control measures for resistant Acinetobacter baumannii and the impact on acquisition of methicillin-resistant Staphylococcus aureus and vancomycin-resistant Enterococcus in a medical intensive care unit. Infect Control Hosp Epidemiol. 2004;25(2):167-8. Epub 2004/03/05. doi: 10.1086/502370. PubMed PMID: 14994945.
- 181. Day HR, Morgan DJ, Himelhoch S, Young A, Perencevich EN. Association between depression and contact precautions in veterans at hospital admission. Am J Infect Control. 2011;39(2):163-5. doi: 10.1016/j.ajic.2010.06.024. PubMed PMID: 21356434; PubMed Central PMCID: PMC3304097.
- 182. Morgan DJ, Diekema DJ, Sepkowitz K, Perencevich EN. Adverse outcomes associated with Contact Precautions: a review of the literature. Am J Infect Control. 2009;37(2):85-93. Epub 2009/03/03. doi: 10.1016/j.ajic.2008.04.257. PubMed PMID: 19249637; PubMed Central PMCID: PMCPMC3557494.
- 183. Abad C, Fearday A, Safdar N. Adverse effects of isolation in hospitalised patients: a systematic review. J Hosp Infect. 2010;76(2):97-102. Epub 2010/07/14. doi: 10.1016/j.jhin.2010.04.027. PubMed PMID: 20619929.
- 184. Siegel JR, E; Jackson, M; Chiarello, L; Heathcare Infection Control Practices Advisory Committee. Management of multidrug-resistant organisms in healthcare settings, 2006. In: Services CfDCaPtDoHaH, editor. 2006.
- 185. Calfee DP, Salgado CD, Classen D, Arias KM, Podgorny K, Anderson DJ, Burstin H, Coffin SE, Dubberke ER, Fraser V, Gerding DN, Griffin FA, Gross P, Kaye KS, Klompas M, Lo E, Marschall J, Mermel LA, Nicolle L, Pegues DA, Perl TM, Saint S, Weinstein RA, Wise R, Yokoe DS. Strategies to prevent transmission of methicillin-resistant Staphylococcus aureus in acute care hospitals. Infect Control Hosp Epidemiol. 2008;29 Suppl 1:S62-80. doi: 10.1086/591061. PubMed PMID: 18840090.
- 186. Huskins WC, Huckabee CM, O'Grady NP, Murray P, Kopetskie H, Zimmer L, Walker ME, Sinkowitz-Cochran RL, Jernigan JA, Samore M, Wallace D, Goldmann DA. Intervention to reduce transmission of resistant bacteria in intensive care. N Engl J Med. 2011;364(15):1407-18. Epub 2011/04/15. doi: 10.1056/NEJMoa1000373. PubMed PMID: 21488763; PubMed Central PMCID: PMCPMC3410743
- 187. Harris AD, Pineles L, Belton B, Johnson JK, Shardell M, Loeb M, Newhouse R, Dembry L, Braun B, Perencevich EN, Hall KK, Morgan DJ, Shahryar SK, Price CS, Gadbaw JJ, Drees M, Kett DH, Munoz-Price LS, Jacob JT, Herwaldt LA, Sulis CA, Yokoe DS, Maragakis L, Lissauer ME, Zervos MJ, Warren DK, Carver RL, Anderson DJ, Calfee DP, Bowling JE, Safdar N. Universal glove and gown use and acquisition of antibiotic-resistant bacteria in the ICU: a randomized trial. JAMA. 2013;310(15):1571-80. Epub 2013/10/08. doi: 10.1001/jama.2013.277815. PubMed PMID: 24097234; PubMed Central PMCID: PMCPMC4026208.

- 188. Safdar N, Marx J, Meyer NA, Maki DG. Effectiveness of preemptive barrier precautions in controlling nosocomial colonization and infection by methicillin-resistant *Staphylococcus aureus* in a burn unit. Am J Infect Control. 2006;34(8):476-83. doi: 10.1016/j.aiic.2006.01.011. PubMed PMID: 17015152.
- 189. Bearman G, Rosato AE, Duane TM, Elam K, Sanogo K, Haner C, Kazlova V, Edmond MB. Trial of universal gloving with emollient-impregnated gloves to promote skin health and prevent the transmission of multidrug-resistant organisms in a surgical intensive care unit. Infect Control Hosp Epidemiol. 2010;31(5):491-7. Epub 2010/03/31. doi: 10.1086/651671. PubMed PMID: 20350197.
- 190. Bearman GM, Marra AR, Sessler CN, Smith WR, Rosato A, Laplante JK, Wenzel RP, Edmond MB. A controlled trial of universal gloving versus contact precautions for preventing the transmission of multidrug resistant organisms. Am J Infect Control. 2007;35(10):650-5. Epub 2007/12/08. doi: 10.1016/j.ajic.2007.02.011. PubMed PMID: 18063129.
- 191. Morgan DJ, Kirkland KB. Uncertainty in the application of contact precautions. Clin Infect Dis. 2012;55(3):474-5. Epub 2012/04/24. doi: 10.1093/cid/cis398. PubMed PMID: 22523270.
- 192. Croft LD, Harris AD, Pineles L, Langenberg P, Shardell M, Fink JC, Simoni-Wastila L, Morgan DJ. The Effect of Universal Glove and Gown Use on Adverse Events in Intensive Care Unit Patients. Clin Infect Dis. 2015. Epub 2015/04/23. doi: 10.1093/cid/civ315. PubMed PMID: 25900169.
- 193. Livorsi DJ, Kundu MG, Batteiger B, Kressel AB. Effect of contact precautions for MRSA on patient satisfaction scores. J Hosp Infect. 2015. Epub 2015/03/24. doi: 10.1016/j.jhin.2015.02.007. PubMed PMID: 25799481.
- 194. Mehrotra P, Croft L, Day HR, Perencevich EN, Pineles L, Harris AD, Weingart SN, Morgan DJ. Effects of contact precautions on patient perception of care and satisfaction: a prospective cohort study. Infect Control Hosp Epidemiol. 2013;34(10):1087-93. Epub 2013/09/11. doi: 10.1086/673143. PubMed PMID: 24018926; PubMed Central PMCID: PMCPMC4070370.
- 195. Day HR, Perencevich EN, Harris AD, Gruber-Baldini AL, Himelhoch SS, Brown CH, Morgan DJ. Depression, anxiety, and moods of hospitalized patients under contact precautions. Infect Control Hosp Epidemiol. 2013;34(3):251-8. Epub 2013/02/08. doi: 10.1086/669526. PubMed PMID: 23388359.
- 196. Day HR, Perencevich EN, Harris AD, Gruber-Baldini AL, Himelhoch SS, Brown CH, Dotter E, Morgan DJ. Association between contact precautions and delirium at a tertiary care center. Infect Control Hosp Epidemiol. 2012;33(1):34-9. doi: 10.1086/663340. PubMed PMID: 22173520; PubMed Central PMCID: PMC3544005.
- 197. Zahar JR, Garrouste-Orgeas M, Vesin A, Schwebel C, Bonadona A, Philippart F, Ara-Somohano C, Misset B, Timsit JF. Impact of contact isolation for multidrug-resistant organisms on the occurrence of medical errors and adverse events. Intensive Care Med. 2013;39(12):2153-60. Epub 2013/09/03. doi: 10.1007/s00134-013-3071-0. PubMed PMID: 23995982.
- 198. Gandra S, Barysauskas CM, Mack DA, Barton B, Finberg R, Ellison RT, 3rd. Impact of contact precautions on falls, pressure ulcers and transmission of MRSA and VRE in hospitalized patients. J Hosp Infect. 2014;88(3):170-6. Epub 2014/12/03. doi: 10.1016/j.jhin.2014.09.003. PubMed PMID: 25441487.
- 199. Lupion-Mendoza C, Antunez-Dominguez MJ, Gonzalez-Fernandez C, Romero-Brioso C, Rodriguez-Bano J. Effects of isolation on patients and staff. Am J Infect Control. 2015;43(4):397-9. Epub 2015/02/28. doi: 10.1016/j.ajic.2015.01.009. PubMed PMID: 25721058.
- 200. Colorado B, Del Toro D, Tarima S. Impact of contact isolation on FIM score change, FIM efficiency score, and length of stay in patients in acute inpatient rehabilitation facility. PM R. 2014;6(11):988-91. Epub 2014/07/06. doi: 10.1016/j.pmrj.2014.05.017. PubMed PMID: 24990448.
- 201. Morgan DJ, Day HR, Harris AD, Furuno JP, Perencevich EN. The impact of Contact Isolation on the quality of inpatient hospital care. PLoS One. 2011;6(7):e22190. Epub 2011/08/04. doi: 10.1371/journal.pone.0022190. PubMed PMID: 21811572; PubMed Central PMCID: PMCPMC3141007.
- 202. Day HR, Perencevich EN, Harris AD, Himelhoch SS, Brown CH, Gruber-Baldini AL, Dotter E, Morgan DJ. Do contact precautions cause depression? A two-year study at a tertiary care medical centre. J Hosp Infect. 2011;79(2):103-7. Epub 2011/06/15. doi: 10.1016/j.jhin.2011.03.026. PubMed PMID: 21664000; PubMed Central PMCID: PMCPMC3331706.
- 203. Morgan DJ, Pineles L, Shardell M, Graham MM, Mohammadi S, Forrest GN, Reisinger HS, Schweizer ML, Perencevich EN. The effect of contact precautions on healthcare worker activity in acute care hospitals. Infect Control Hosp Epidemiol. 2013;34(1):69-73. doi: 10.1086/668775. PubMed PMID: 23221195.
- 204. Huang SS, Septimus E, Kleinman K, Moody J, Hickok J, Avery TR, Lankiewicz J, Gombosev A, Terpstra L, Hartford F, Hayden MK, Jernigan JA, Weinstein RA, Fraser VJ, Haffenreffer K, Cui E, Kaganov RE, Lolans K, Perlin JB, Platt R, Program CDCPE, Network AD, Healthcare-Associated Infections P. Targeted versus universal decolonization to prevent ICU infection. N Engl J Med. 2013;368(24):2255-65. doi: 10.1056/NEJMoa1207290. PubMed PMID: 23718152.
- 205. Schweizer M, Perencevich E, McDanel J, Carson J, Formanek M, Hafner J, Braun B, Herwaldt L. Effectiveness of a bundled intervention of decolonization and prophylaxis to decrease Gram positive surgical site infections after cardiac or orthopedic surgery: systematic review and meta-analysis. BMJ. 2013;346:f2743. doi: 10.1136/bmj.f2743. PubMed PMID: 23766464; PubMed Central PMCID: PMC3681273.
- 206. Feazel LM, Malhotra A, Perencevich EN, Kaboli P, Diekema DJ, Schweizer ML. Effect of antibiotic stewardship programmes on Clostridium difficile incidence: a systematic review and meta-analysis. J Antimicrob Chemother. 2014;69(7):1748-54. Epub 2014/03/19. doi: 10.1093/jac/dku046. PubMed PMID: 24633207.
- 207. Formanek MB, Herwaldt LA, Perencevich EN, Schweizer ML. Gentamicin/collagen sponge use may reduce the risk of surgical site infections for patients undergoing cardiac operations: a meta-analysis. Surg Infect (Larchmt). 2014;15(3):244-55. Epub 2014/04/30. doi: 10.1089/sur.2012.209. PubMed PMID: 24773201; PubMed Central PMCID: PMCPMC4063378.
- 208. Schweizer ML, Reisinger HS, Ohl M, Formanek MB, Blevins A, Ward MA, Perencevich EN. Searching for an optimal hand hygiene bundle: a meta-analysis. Clin Infect Dis. 2014;58(2):248-59. Epub 2013/10/11. doi: 10.1093/cid/cit670. PubMed PMID: 24107409. 209. Nair R, Ammann E, Rysavy M, Schweizer ML. Mortality among patients with methicillin-resistant Staphylococcus aureus USA300 versus non-USA300 invasive infections: a meta-analysis. Infect Control Hosp Epidemiol. 2014;35(1):31-41. Epub 2013/12/18. doi: 10.1086/674385. PubMed PMID: 24334796.

- 210. Schweizer ML, Bossen A, McDanel JS, Dennis LK. Staphylococcus aureus colonization before infection is not associated with mortality among S. aureus-infected patients: a meta-analysis. Infect Control Hosp Epidemiol. 2012;33(8):796-802. Epub 2012/07/05. doi: 10.1086/666628. PubMed PMID: 22759547.
- 211. 2014 Ebola Outbreak in West Africa Case Counts: Centers for Disease Control and Prevention; [May 20, 2015]. Available from: http://www.cdc.gov/vhf/ebola/outbreaks/2014-west-africa/case-counts.html.
- 212. Cochrane Handbook for Systematic Reviews of Interventions: The Cochrane Collaboration; 2011. Available from: www.cochrane-handbook.org.
- 213. Stroup DF, Berlin JA, Morton SC, Olkin I, Williamson GD, Rennie D, Moher D, Becker BJ, Sipe TA, Thacker SB. Meta-analysis of observational studies in epidemiology: a proposal for reporting. Meta-analysis Of Observational Studies in Epidemiology (MOOSE) group. JAMA. 2000;283(15):2008-12. Epub 2000/05/02. PubMed PMID: 10789670.
- 214. Liberati A, Altman DG, Tetzlaff J, Mulrow C, Gotzsche PC, Ioannidis JP, Clarke M, Devereaux PJ, Kleijnen J, Moher D. The PRISMA statement for reporting systematic reviews and meta-analyses of studies that evaluate healthcare interventions: explanation and elaboration. BMJ. 2009;339:b2700. Epub 2009/07/23. doi: 10.1136/bmj.b2700. PubMed PMID: 19622552; PubMed Central PMCID: PMCPMC2714672.
- 215. Stang A. Critical evaluation of the Newcastle-Ottawa scale for the assessment of the quality of nonrandomized studies in meta-analyses. Eur J Epidemiol. 2010;25(9):603-5. Epub 2010/07/24. doi: 10.1007/s10654-010-9491-z. PubMed PMID: 20652370.
- 216. N DRL. Fixed and Random Effects Models: Meta-analysis in clinical trials. Controlled Clinical Trials. 1986;7:177-88.
- 217. Review Manager (RevMan). Version 5.3 ed. Copenhagen: The Nordic Cochrane Center, The Cochrane Collaboration; 2011.
- 218. Kennedy P, Hamilton LR. Psychological impact of the management of methicillin-resistant Staphylococcus aureus (MRSA) in patients with spinal cord injury. Spinal Cord. 1997;35(9):617-9. Epub 1997/09/25. PubMed PMID: 9300970.
- 219. Catalano G, Houston SH, Catalano MC, Butera AS, Jennings SM, Hakala SM, Burrows SL, Hickey MG, Duss CV, Skelton DN, Laliotis GJ. Anxiety and depression in hospitalized patients in resistant organism isolation. South Med J. 2003;96(2):141-5. Epub 2003/03/13. doi: 10.1097/01.smj.0000050683.36014.2e. PubMed PMID: 12630637.
- 220. Petitti DB. Meta-Analysis, Decision Analysis, and Cost-Effectiveness Analysis: Methods for Quantitative Synthesis in Medicine. 2nd ed. New York: Oxford University Press; 2000.
- 221. Chan KY, Wang W, Wu JJ, Liu L, Theodoratou E, Car J, Middleton L, Russ TC, Deary IJ, Campbell H, Wang W, Rudan I. Epidemiology of Alzheimer's disease and other forms of dementia in China, 1990-2010: a systematic review and analysis. Lancet. 2013;381(9882):2016-23. Epub 2013/06/12. doi: 10.1016/s0140-6736(13)60221-4. PubMed PMID: 23746902.
- 222. Harbord RM, Egger M, Sterne JA. A modified test for small-study effects in meta-analyses of controlled trials with binary endpoints. Stat Med. 2006;25(20):3443-57. Epub 2005/12/14. doi: 10.1002/sim.2380. PubMed PMID: 16345038.

#### 1.3 Risks

The risks to participants are minimal. There is a risk the Provodine $^{TM}$  may cause very mild skin irritation. In addition, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study. Hand cultures collected from participants will be labelled with a study number.

## 1.4 Benefits

There are no direct benefits to participants from being in this study. However, we hope that, in the future, other people might benefit from this study because this study may help us identify ways to decrease self-contamination while removing personal protective equipment and, thereby, possibly decrease the risk of transmission of infectious diseases from patient to healthcare worker.

### 1.5 Risk Benefit Ratio

The potential benefits of this study outweigh the minimal risks to participants.

## 2 Study Objectives, Aims, and Hypothesis

Participants will serve as their own controls in this pilot study, first in a control arm then a ProvodineTM arm.

Hypothesis: We hypothesize that Provodine<sup>™</sup> will protect participants' hands from contamination with the test contaminants during PPE removal. Bacterial growth from the bag-broth cultures from the Provodine<sup>™</sup> arm will have significantly less growth than from the control arm.

## 3 Study Design and Procedure

Study Design: We will perform a two-armed pilot test among 40 front-line healthcare workers (nurses, doctors, respiratory therapists, etc) at the University of Iowa Hospitals and Clinics. Participants will serve as their own controls. First, participants will perform hand hygiene with alcohol-based hand rub as they normally would in clinical practice then don PPE. We, the research team, will contaminate participating healthcare workers' (HCW) PPE with either bacteriophage MS2 (twenty participants) or S. marcescens ATCC 14756 (twenty participants). MS2 preparation and propagation and S. marcescens culture suspensions will each be performed as previously described. (123, 124) The MS2 bacteriophage will be suspended in 0.01 M phosphate-buffered saline and each PPE site will be contaminated with 105 plaque-forming units (PFU) of MS2 in 5 drops of 5 µL each. Aliquots of 3 mL of S. marcescens broth suspension (yielding bacterial titers of ~1 X 109 CFU/ml) will be applied to each PPE site. Participants will then doff PPE using the Centers for Disease Control's (CDC) recommended protocol. We will sample their hands using the bag broth method. A research assistant will monitor participants as they wash their hands with soap and water then rinse their hands with 70% ethanol. Participants will then apply Provodine<sup>TM</sup> to their hands and put on (don) fresh PPE. We will repeat the contamination, doffing, and sampling procedure. For MS2 recovery, we will assay the eluent using the most probable number (MPN) enrichment infectivity assay.(126) For S. marcescens recovery, we will dilute the eluent, plate it, incubate the plates, and count the colonies as described.(124, 127)

## 4 Selection and Withdrawal of Participants

### 4.1 Selection of Study Population

Email, plus referral from colleague? Nurses, doctors, others?

### 4.2 Inclusion Criteria

Front-line healthcare workers (how to make sure we get clinical staff who use PPE regularly?)

#### 4.3 Exclusion Criteria

Healthcare workers with known skin allergies to povidone iodine.

## 4.4 Participant Withdrawal

Participants may withdraw from the study at any time. Any cultures collected from participants wishing to withdraw will be destroyed.

#### 4.5 Participant Compensation

Upon completion of the two study arms, participants will receive a \$30 gift card to thank them for their time. Gift cards will be sent from the XXXXXX to participants via University of Iowa Campus Mail.

#### 5 Informed Consent Process

#### 5.1 Recruitment

Email? Referral?

Then set up appointment for consent – where will we do this? Lab?

# 5.2 Informed Consent Process

Participant meet with RA, go through consent form, questions, proceed immediately to pilot test. Whole thing take 2 hours?

### 6 Statistical Plan

#### 6.1 Power Calculations

On the basis of the literature, we assumed that 80%-90% of participants will contaminate themselves with MS2 and 60%-70% with S. marcescens. If Provodine<sup>TM</sup> is effective, 20 participants in each group would provide 80% power to detect a 60%-70% relative decrease (rate ratio = 0.3 to 0.4) in the rate of self-contamination (present or absent) and higher power to find a significant difference in the quantity of MS2 or S. marcescens recovered from participants' hands.

## 6.2 Analytical Plan

We will use the paired t-test or Wilcoxon signed-rank test to compare the quantity of MS2 bacteriophage or S. marcescens recovered after participants who applied Provodine<sup>TM</sup> to their hands before donning gloves with the quantity recovered from the control arm where participants who did hand hygiene with an alcohol-based product before donning gloves.

### 7 Data Collection, Handling, and Storage

All data collected will be stored in an electronic database on a shared drive within the University of Iowa Healthcare servers. Only members of the research team will have access to the database. No PHI will be collected. All participants will be identified in the database by a study number.

We will bank the isolates so that we can do susceptibility testing and pulsed field gel electrophoresis (PFGE) on the isolates in the future if this information is deemed important. All cultures and isolates will be labelled with study numbers and stored in XXXXXXXXX in the Diekema lab.